CLINICAL TRIAL: NCT04444609
Title: PROSAIC-19 - Prospective Longitudinal Assessment in a COVID-19 Infected Cohort
Acronym: PROSAIC-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20IC5943
Record Dates: First submitted 2020-06-16; First posted 2020-06-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; SARS-CoV 2; ARDS, Human; Immune System Disorder
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Immune System Diseases | interventions — Nasal Lavage; Toothbrushing; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spontaneously expectorated sputum, nasal lavage, brushings and nasal synthetic absorptive matrix (SAM) samples
  Venous blood (60mls) will be taken into Lithium Heparin tubes and PAXgene RNA tubes
  PAXgene tubes will be stored at -80C for further host genetic sequencing analysis. Further immunological analysis using yeast surface display for serum antibody profiling, single B cell sorting to generate monoclonal antibodies and ELISPOT to analyse CD4 and CD8 T cell ELISPOT to SARS CoV-2 peptide pools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- COVID -19 with chronic lung disease: Subjects with swab confirmed COVID-19 and underlying chronic lung disease (n=60)
  Severe (n=30) (defined by presence of ARDS, sepsis or severe pneumonia)
  Mild/Moderate ( n =30) (absence of severe criteria)
  Interventions: Other: Blood tests sputum, nasal lavage and brushing
- COVID-19 without chronic lung disease: Subjects with swab confirmed COVID-19 and no chronic lung disease (n=60)
  Severe (n=30) (defined by presence of ARDS, sepsis or severe pneumonia)
  Mild/Moderate ( n =30) (absence of severe criteria)
  Interventions: Other: Blood tests sputum, nasal lavage and brushing
- Chronic Lung disease: Subjects with chronic lung disease (identified as requiring shielding based on severity) but no COVID-19 (n=80)
  * Asthma (defined as severe) - (n=20)
  * CF (FEV1% predicted baseline <50%) - (n=20)
  * COPD (FEV1% predicted baseline <50%) - (n=20)
  * Idiopathic Pulmonary Fibrosis (n=20)
  Interventions: Other: Blood tests sputum, nasal lavage and brushing
- Healthy volunteers: Healthy subjects with no COVID-19 (n=30)
  Interventions: Other: Blood tests sputum, nasal lavage and brushing

INTERVENTIONS:
Other: Blood tests sputum, nasal lavage and brushing — Venesection, sputum nasal lavage and brushing if appropriate
  Other Names: Blood tests; Sputum; Nasal lavage; Nasal brushings; EndoPAT

SUMMARY:
DESIGN Longitudinal prospective observational multicentre study.

Primary objective:

Understand the immune mechanisms driving COVID-19 disease in patients with a history of lung disease

DETAILED DESCRIPTION:
INTRODUCTION

1.1 BACKGROUND

Coronavirus disease 2019 (COVID-19) caused by SARS-CoV-2 infection is a new rapidly spreading infectious disease with no proven treatment options. The virus causes a spectrum of disease ranging from mild coryzal symptoms to severe respiratory compromise requiring ventilatory support. Guidance from Public Health England identifies several groups that are at risk of severe disease including the elderly and individuals with chronic lung disease. Additionally, there is also debate over the role of corticosteroids with some hospital guidelines recommending their use despite WHO guidance contradicting this due to concerns that they may impair antiviral immunity and worsen disease. The mechanisms driving severity of disease in certain individuals infected with COVID-19 are poorly understood. We urgently need to understand these mechanisms to facilitate rapid development of novel effective therapies and vaccines

1. Immunosusceptibility to severe COVID-19 disease

There are several putative mechanisms through which SARS-CoV-2 could drive greater disease severity in pre-disposed individuals. These include:

1. Impaired innate anti-viral immune responses

   Following viral entry, the innate immune response to respiratory viruses involves induction of the type I and III interferons (IFN). This initiates a cascade that triggers expression of a range of interferon-stimulated genes expressing proteins that act in concert to limit viral replication. Chronic lung diseases, particularly asthma, cystic Fibrosis (CF) and COPD are associated with impaired or dysregulated induction of interferon to commonly encountered viruses such as rhinovirus and influenza and similar dysregulation may occur with SARS-CoV-2. Inhaled interferon-β is currently in trials as an anti-viral therapy for asthma and COPD.
2. Exaggerated inflammatory responses to viral infection

   Common respiratory viral infections such as influenza and respiratory syncyitial virus (RSV) can promote viral pathology mediated by antibodies and T cell responses. Early evidence suggests that severe COVID-19 disease is associated with hyperinflammation, a feature that could be directly driven by virus burden or occur due to independent hyperactivation of the immune system. Human coronavirus infections including SARS-CoV can induce immunopathology in the lungs through a number of different mechanisms including antibody enhancement of SARS-CoV infection by human macrophages. Significant increases in CD4 and CD8 expressing pro-inflammatory cytokines have been shown in severe SARS-CoV disease compared to mild/moderate disease.

   Accordingly, there has been considerable interest in a potential role of repurposing existing immunosuppressive therapies for treatment of severe COVID-19. The key mediators and pathways that drive hyperinflammation in COVID-19 are unclear and greater elucidation of these processes will inform repurposing of existing therapies or development of novel approaches to effective treatment. The implication of baseline dysregulated T cell responses such as those seen in chronic lung disease (e.g. asthma, COPD, Cystic Fibrosis) is again unclear and requires further mechanistic understanding. As such it is, as yet, unclear whether immunosuppressive therapies currently in clinical trials will be beneficial or harmful in these large cohorts of susceptible patients.
3. Dysregulated interferon-dependent endothelial function to COVID-19

   Acute respiratory distress syndrome (ARDS) is characterised by hydrostatic pulmonary oedema, elevated pulmonary vascular resistance and coagulopathy, there is disruption of endothelial function with dysregulated release of the endothelially derived vasoactive hormones. Circulating levels of endothelin-1 are raised in patients with ARDS[16], likely due to increased production and decreased clearance in the lungs potentially regulated by Angiopoietin-1.

   Severe SARS-CoV-2 infection is associated with cytokine storm. Raised serum levels of a number of key inflammatory cytokines including IFN-gamma, TNF-alpha, IP10, IL-8 and IL-10 and elevated levels of IL-6 are strongly associated with mortality. IL-6 release is synergistically induced by IFN-gamma and TNF-alpha and in a positive feedback mechanism, a low dose of IL-6 strongly enhances the cellular responses to IFN-alpha and modulates interferon-stimulated gene expression. In an experimental murine model, we found that infection with rhinovirus with IFN co-stimulation leads to elevated bronchoalveolar lavage levels of IL-6 (Singanayagam et al, unpublished observations). These data suggest that in patients with severe COVID-19, a hyperinflammatory process ensues and we hypothesise that through dysregulated and unchecked IFN production, key vasculo-inflammatory interferon-stimulated genes including IP10 and ET-1 drive worse outcomes with increased parenchymal and pulmonary vascular inflammation. This results in a dichotomy whereby initial IFN induction is required to limit viral replication, but late unchecked production can worsen pathophysiology. This is supported by emerging clinical data suggesting a unique phenotype to SARS-CoV-2 critical care patients characterised by severe hypoxia with near normal lung compliance.
4. Altered viral entry receptor expression: Recent data indicates SARS-CoV-2 utilises angiotensin-converting enzyme (ACE)2 as a receptor for viral attachment and also the protease TMPRSS2 which cleaves the spike(S) protein to allow fusion of the virus with cellular membranes. ACE2 and TMPRSS2 are frequently co-expressed in the pulmonary epithelium. A recent study also showed that ACE2 is an interferon stimulated gene (ISG)(i.e. directly induced by the anti-viral response) and therefore, SARS-CoV-2 might upregulate its own receptor to propagate infection. Recent data indicates that smokers and subjects with chronic obstructive pulmonary disease (COPD) have increased pulmonary ACE2 expression suggesting that chronic lung disease might facilitate greater infection with SARS-CoV-2. Conversely, ACE2 expression protects against acute lung injury in the context of acid aspiration or sepsis and therefore, if ACE2 induction by SARS-CoVs is impaired in chronic lung disease, this could predispose to adverse outcome.
5. Increased secondary bacterial and/or fungal infections

In early case series, secondary infections have been observed more frequently in subjects with severe COVID-19 disease. Secondary bacterial infection is a well-recognised phenomenon following rhinovirus, influenza or respiratory syncytial virus and may be mechanistically driven by a range of possible mechanisms including macrophage phagocytosis or neutrophil elastase-mediated cleavage of anti-microbial peptides. These processes may be worsened by use of corticosteroids28 and, notably, a greater proportion of patients with secondary infections following COVID-19 had been prescribed steroids.

Invasive fungal disease consistent with aspergillosis has also been observed for both severe acute respiratory syndrome coronavirus (SARS-CoV-2003) and Middle East Respiratory Syndrome coronavirus (MERS-CoV), and anecdotal reports of post-mortems in patients with COVID-19 from China suggest that Aspergillus pulmonary infections occur. These data are early warning signs that secondary invasive fungal infections may present an increasingly serious complication in patients affected with COVID-19 as the pandemic progresses. Understanding the mechanistic basis for immune susceptibility to secondary bacterial/fungal infection and an ability to prevent these secondary infections could be a key step towards improving outcomes from the disease.

1.2 RATIONALE FOR CURRENT STUDY

In this study, the investigators will analyse blood and airway samples from individuals with confirmed COVID-19 to understand the immune mechanisms that lead to severe disease. We will elucidate specific mechanisms that drive more severe pathology in higher risk individuals such as those with chronic lung disease. Through detailed immunoprofiling, we will identify key pathways and druggable targets to exploit in future clinical intervention studies.

Hypotheses:

1. High risk individuals including individuals with chronic lung disease have impaired anti-viral immune responses to SARS-CoV-2, increasing virus-induced inflammation.
2. Interferon-dependent endothelial dysfunction drives pathogenicity in SARS-CoV-2 infection.
3. Susceptibility to secondary bacterial and fungal infection in chronic lung disease is related to selective pathway defects in innate immune function.

2. STUDY OBJECTIVES

Primary objective:

1. Understand the immune mechanisms driving COVID-19 disease in patients with a history of lung disease

Secondary objectives

1. Identify immune correlates of protection and lung pathology in SARS-CoV-2 infection.
2. Analysis of endothelial function in mild and severe COVID-19 patients and ex vivo using virus stimulated blood-derived endothelial cells from patients with COVID-19.
3. Evaluation of changes in upper/lower airway microbiota and mycobiota occurring during COVID-19.
4. Evaluation of ex vivo peripheral blood immune responses to viral, bacterial and fungal stimuli in patients with COVID-19 and chronic lung disease in comparison to patients with COVID-19 and no chronic lung disease.
5. Analysis of quality of life impact of COVID-19 infection in chronic lung disease.

3. STUDY DESIGN

Through a 24 month prospective longitudinal multicentre (Royal Brompton & Harefield NHS Trust Chelsea and Westminster NHS Foundation Trust, and Imperial College Healthcare NHS Trusts) observational study, the study team will analyse blood, sputum and nasal sampling alongside non-invasive EndoPAT device testing in a total pf 230 subjects. The study team will obtain peripheral blood, sputum, nasal lavage, brushings and nasal synthetic absorptive matrix (SAM) samples and perform non-invasive EndoPAT testing on the day of hospital presentation and at weekly intervals during inpatient setting and then during outpatient visits post-discharge over a 12 month follow-up period. The study team will collect clinical information including demographics, routine laboratory investigations, clinical symptom scores and outcomes. Linked pseudoanonymised radiology imaging will also be transferred for analysis.

Spontaneously expectorated sputum, nasal lavage, brushings and nasal synthetic absorptive matrix (SAM) samples will be taken and processed as previously described and stored at -800C for downstream analyses including ELISA/MSD, viral load measurement and microbiome analysis. Venous blood (60mls) will be taken into Lithium Heparin tubes and PAXgene RNA tubes and transferred to Imperial College (RBH) for processing and storage. PBMCs will be extracted for in vitro stimulation assays and whole blood (1ml) and serum (2mls) isolated and stored at -80oC for further analysis. PAXgene tubes will be stored at -80C for further host genetic sequencing analysis. Further immunological analysis using yeast surface display for serum antibody profiling, single B cell sorting to generate monoclonal antibodies and ELISPOT to analyse CD4 and CD8 T cell ELISPOT to SARS CoV-2 peptide pools. Further deep immunological profiling using cytokine analysis, PBMC cytokine response to viral (or viral PRR agonist), fungal stimuli, yeast surface display for serum antibody profiling, single memory B cell expression cloning will be carried. CD4 and CD8 T cell ELISPOT will be performed as previously described. Non-invasive EndoPAT testing will also be performed as previously described.

ELIGIBILITY:
Inclusion Criteria:

1. All patients ≥16 years old with confirmation of COVID-19
2. All patients ≥ 16 years old with chronic lung disease (CF, non-CF bronchiectasis, asthma, COPD or Idiopathic Pulmonary Fibrosis) or with no evidence of prior chronic lung disease
3. Healthy volunteers

Exclusion Criteria:

None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with swab confirmed COVID-19 and underlying chronic lung disease (n=60)
  * Severe (n=30) (defined by presence of ARDS, sepsis or severe pneumonia)
  * Mild/Moderate ( n =30) Absence of features of severe disease
  Subjects with swab confirmed COVID-19 and no chronic lung disease (n=60)
  * Severe (n=30) (defined by presence of ARDS, sepsis or severe pneumonia)
  * Mild/Moderate ( n =30) Absence of features of severe disease
  Subjects with chronic lung disease (identified as requiring shielding based on severity) but no COVID-19 (n=80)
  * Asthma (defined as severe) - (n=20)
  * CF (FEV1% predicted baseline <50%) - (n=20)
  * COPD (FEV1% predicted baseline <50%) - (n=20)
  * Idiopathic Pulmonary Fibrosis (n=20)
    3.Healthy subjects with no COVID-19 (n=30)
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Anti-viral cytokine levels in blood samples in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Anti-viral cytokine protein concentration in blood samples by ELISA
Anti-viral cytokines profiles within sputum samples in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Inflammatory cytokine protein concentration in sputum samples by ELISA
Anti-viral cytokine profiles within nasal lavage samples in chronic respiratory disease associated with susceptibility to severe COVID-19 infection associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Inflammatory cytokine protein concentration in nasal lavage samples by ELISA
Expression of inflammatory gene expression in upper respiratory epithelial airway cells using nasal brush specimens in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Inflammatory gene expression in upper airway respiratory epithelial cells by RNA sequencing.

SECONDARY OUTCOMES:
Identify the T cell antigens and B cell epitopes in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Analysis of viral components recognized by the adaptive immune system
Peripheral blood mononuclear cell (PBMC) interferon mediated immune responses to pathogen recognition receptor agonists in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Cytokine protein concentration following PBMC stimulation to pathogen recognition receptor agonists by Elispot
Identify endothelial function in chronic respiratory disease associated with susceptibility to severe COVID-19 infection using EndoPAT testing | Through study completion an average of 1 year
  Analysis of endothelial function
Endothelial cell inflammation biomarkers in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Serum and plasma protein concentration of endothelial cell inflammation biomarkers by ELISA
Identify sputum 16S rRNA and ITS sequences in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Analysis of sputum microbiome
Identify nasal lavage 16S rRNA and ITS sequences in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Analysis of nasal microbiome
Identify quality of life markers in chronic respiratory disease associated with susceptibility to severe COVID-19 infection | Through study completion an average of 1 year
  Study participant survey

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kelleher, MD PhD, Study Chair — Imperial College London
Locations (1):
- Royal Brompton & Harefileld NHS Trusts, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Under consideration